CLINICAL TRIAL: NCT04025528
Title: Pathophysiology of Hypoventilation in Obesity and Effects of Bariatric Intervention: PHOEBI Study
Brief Title: Pathophysiology of Hypoventilation in Obesity and Effects of Bariatric Intervention
Acronym: PHOEBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 258045
Record Dates: First submitted 2019-06-21; First posted 2019-07-19 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Obesity Hypoventilation Syndrome (OHS)
MeSH Terms: conditions — Obesity Hypoventilation Syndrome | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypercapnic: Obese patients with daytime hypercapnia
  Interventions: Procedure: Bariatric Surgery
- Eucapnic: Obese patients with normal daytime carbon dioxide levels
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — Weight loss surgery with either gastric sleeve or gastric bypass surgery

SUMMARY:
Breathing is impacted by obesity. Early changes are characterised by significant breathing abnormalities during sleep (a condition called sleep disordered breathing, the most common of which is obstructive sleep apnoea). As the breathing changes worsen in severity, it may result in a rise in carbon dioxide levels during daytime causing a condition called obesity hypoventilation syndrome (OHS). The current treatment for obesity related breathing changes include supportive breathing therapy at night, optimisation of associated medical conditions and weight loss.

Weight management is an important part of obesity treatment. Weight loss strategies such as life-style modification do not always work. Weight loss surgery (bariatric surgery) has been shown to be an effective weight management intervention with long-term results. This study aims to understand breathing changes that occurs due to obesity and their resolution after weight loss surgery. The investigators are aiming to recruit participants with sleep disordered breathing who are currently awaiting bariatric surgery. In particular, the investigators are interested in comparing breathing changes in participants with OHS, who have abnormal regulation of their carbon dioxide levels, and participants with sleep disordered breathing with normal CO2 regulation.

Participants will be recruited through outpatient clinics for sleep disordered breathing. The participants will undergo comprehensive breathing assessments on enrolment including an overnight sleep study. Participants will undergo further daytime breathing assessments before and after their bariatric surgery. End of study will be 6 months after surgery - participants will have a final comprehensive breathing assessment including an overnight sleep study to review resolution of their breathing changes. Depending on the wait list time for the bariatric surgery, it is anticipated that participants will be enrolled in the study for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older
2. BMI > 40
3. Patients with significant sleep disordered breathing requiring treatment
4. Patient is being assessed for bariatric surgery for either gastric sleeve or gastric bypass surgery

Exclusion Criteria:

1. Patients with decompensated hypercapnic respiratory failure (pH< 7.3)
2. Chronic hypercapnic respiratory failure due to a cause other than obesity such as neuromuscular, chest wall or airway disease
3. Unstable cardiac disease including coronary artery disease and heart failure
4. Significant co-morbid psychiatric disease requiring anti-psychotic medications
5. Chronic pain syndrome on high dose opioid medications
6. Treatment for drug or alcohol addiction
7. Cognitive impairment that would prevent informed consent
8. Pregnancy
9. Need for long-term renal replacement therapy
10. Patients who undergo bariatric intervention with gastric balloon or gastric band.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese patients who are considering bariatric surgery intervention
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Expiratory flow limitation as measured by forced oscillation testing | Measurements on enrolment into study; measurements prior to bariatric surgery (once patients has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Measurement of expiratory flow limitation at different position including upright, 45 degrees and supine. We will explore whether expiratory flow limitation can differentiate hypercapnic and eucapnic patients
Degree of change in expiratory flow limitation | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Explore whether the degree of positional change in expiratory flow limitation can differentiate between eucapnic and hypercapnic patients

SECONDARY OUTCOMES:
Closing capacity | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Measurement of closing capacity at different position including upright, 45 degrees and supine. We will explore whether expiratory flow limitation can differentiate hypercapnic and eucapnic patients
Degree of change in closing capacity | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Explore whether the degree of positional change in closing capacity can differentiate between eucapnic and hypercapnic patients
Correlation between closing capacity and expiratory flow limitation | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Compare outcome 1 and 3 to explore whether there is a relationship between expiratory flow limitation and closing capacity
Intra-abdominal pressure | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  We will measure intra-abdominal pressure and explore whether hypercapnic patients have increased intra-abdominal pressure. Positional changes will be measured
Correlation between intra-abdominal pressure, closing capacity and expriatory flow limitation | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Compare outcome 1,3 and 6. This is a complex multi-compartment model that can differentiate hypercapnia and eucapnic patients
Upper airway collapsibility | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Measurement of upper airway collapsibility as measure by negative expiratory pressure. Explore whether there is a relationship between hypercapnic and eucapnic patients depending on degree of upper airway collapsibility
Lung compliance | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Measurement of lung compliance with pressure volume curve including measurements in different positions (upright, 45 degrees and supine)
Respiratory muscle strength (maximal inspiratory pressure/maximal expiratory) | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Measurement of inspiratory and expiratory muscle strength
Respiratory muscle strength (SNIP test) | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Measurement of sniff nasal inspiratory pressure
Daytime neural respiratory drive (para-sternal electromyography measurements) | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Daytime neural respiratory drive as measured by parasternal electromyography (EMG) measurements can differentiate between hypercapnic and eucapnic patients
Daytime neural respiratory drive (diaphragm electromyography measurements) | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Daytime neural respiratory drive as measured by diaphragm electromyography (EMG) measurements can differentiate between hypercapnic and eucapnic patients
Nocturnal neural respiratory drive (para-sternal electromyography measurements) | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Nocturnal neural respiratory drive as measured by parasternal electromyography (EMG) measurements can differentiate between hypercapnic and eucapnic patients
Nocturnal neural respiratory drive (diaphragm electromyography measurements) | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Nocturnal neural respiratory drive as measured by diaphragm electromyography (EMG) measurements can differentiate between hypercapnic and eucapnic patients
Quality of life post bariatric surgery with SF-36 | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Quality of life changes after bariatric surgery more than with standard medical therapy
Quality of life post bariatric surgery with EQ-5D | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Quality of life changes after bariatric surgery more than with standard medical therapy
Symptom change after commencement of medical therapy compared to bariatric surgery measured with Epworth Sleepiness Scale | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Symptom change after bariatric surgery is more than with standard medical therapy
Symptom change after commencement of medical therapy compared to bariatric surgery measured with mMRC (modified medical research council) dypnoea score | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Symptom change after bariatric surgery is more than with standard medical therapy
Symptom change after commencement of medical therapy compared to bariatric surgery measured with Multi-dimensional dyspnoea profile | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Symptom change after bariatric surgery is more than with standard medical therapy
Symptom change after commencement of medical therapy compared to bariatric surgery measured with Severe Respiratory Insufficiency Questionnaire | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Symptom change after bariatric surgery is more than with standard medical therapy
Changes in healthcare resource usage in OHS patients post bariatric surgery | 6 months pre bariatric surgery and 6 months post bariatric surgery
  Estimation of healthcare usage cost in the 6 months prior to surgery and 6 months post surgery including medication costs and re-admissions to hospital
Improvement in daytime CO2 levels | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Arterial blood gas performed before and after bariatric surgery with improvement in CO2 levels
Improvement in apnoea-hyponoea index | Before bariatric surgery on enrolment and 6 months after bariatric surgery
  Patients will have diagnostic sleep study before and after bariatric surgery
Improvement in mean nocturnal oxygen saturation during sleep | Before bariatric surgery on enrolment and 6 months after bariatric surgery
  Patients will have diagnostic sleep study before and after bariatric surgery
Improvement in mean time spent below 90% oxygen saturation during sleep | Before bariatric surgery on enrolment and 6 months after bariatric surgery
  Patients will have diagnostic sleep study before and after bariatric surgery
Changes in sleep architecture measured by %slow wave sleep and %REM sleep | Before bariatric surgery on enrolment and 6 months after bariatric surgery
  Patients will have diagnostic sleep study before and after bariatric surgery
Improvement in diaphragm function | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  Diaphragm thickening will be measured by ultrasound assessment
Improvement in glycaemic control | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  HbA1C will be measured before and after bariatric surgery

OTHER OUTCOMES:
Spectrum of sleep disordered breathing | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  We will look at sub-group analyses for outcomes 1-29 based on degree of hypoventilation as defined by ERS/ESRS working group
Choice of bariatric surgery | Measurements on enrolment into study; measurements prior to bariatric surgery (once patient has a surgery date); measurements 2-4 weeks after bariatric surgery; and end of study measurements 6 months after bariatric surgery
  We will investigate whether outcomes 1-29 is different depending on type of surgery the patient undergoes (gastric bypass compared to gastric sleeve)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Steier, PhD, Principal Investigator — Guy's and St Thomas NHS Trust
Locations (1):
- Guy's and St Thomas' NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided